CLINICAL TRIAL: NCT05722860
Title: Effect of Oral L-Citrulline on the Peripheral and Central Endothelial Function in Young and Older Adults
Brief Title: L-Citrulline and Endothelial Function
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15485
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Aging
Keywords: L-Citrulline
MeSH Terms: interventions — Citrulline; Capsules

STUDY DESIGN:
Intervention Model Description: Open label single arm study
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- L-Citrulline (Experimental): L-Citrulline 50 g/day per os for 1 week
  Interventions: Drug: L-Citrulline, capsule

INTERVENTIONS:
Drug: L-Citrulline, capsule — 5g/daily dose for the duration of 1 week intervention

SUMMARY:
The effect of L-Citrulline is well studied in relation to muscle strength, exhaustion, exercise performance, and endothelial function in health and disease. This study will extend current body of knowledge and will investigate the effect of L-Citrulline on brain vascular function.

DETAILED DESCRIPTION:
Endothelial function is associated with nitric oxide (NO) availability for vasodilation, blood pressure and blood flow regulation, and vascular health. A large body of evidence demonstrates that aging is associated with a decrease in bioavailability of NO, with more pronounced decrease in sedentary individuals. NO can be produced via the NO synthase (NOS) enzymes, which catalyze the conversion of L-Arginine - a semi-essential amino acid found in fish, nuts and legumes amongst others - to L-Citrulline and produce NO as an endproduct. While the effect of L-Citrulline is extensively studied in relation to muscle strength, exhaustion, exercise performance, as well as on endothelial function in healthy and diseased individuals (including obese and those with heart failure), the effect of L-Citrulline on brain vascular function is not well studied.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-45 and ≥55-90 years of age
* Adequate hearing and visual acuity to participate in the examinations
* Ability to read and write in English
* Competence to provide informed consent

Exclusion Criteria:

* Active CNS disease including multiple sclerosis, uncontrolled seizures, active brain cancer
* Cerebrovascular accident other than TIA within 60 days prior to Visit 0
* Major psychiatric disease, including major depression not currently controlled on medications, alcohol or drug abuse
* Treatment with other Citrulline enhancers (L-Arginine, L-Citrulline Malate) within 4 weeks prior to Visit 0
* Any other medical condition which, in the opinion of investigator, would render the patient inappropriate or too unstable to complete the study protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Change in neurovascular coupling using functional near infrared spectroscopy (fNIRS) | 1 week
  Functional near infrared spectroscopy (fNIRS) will be performed during the cognitive n-back task. fNIRS approach generates data that represent a relative change in oxygenated and deoxygenated hemoglobin measured over the cortical brain tissues. Neurovascular coupling will be evaluated as a change in oxy- and deoxy-hemoglobin between before and after treatment. Units of measure - beta. Reported as a %change from baseline, before and after treatment.
Change in neurovascular coupling using the dynamic retinal vessel analysis | 1 week
  Flicker light-induced dilation of the retinal vessels (percentage increase over baseline diameter) will be measured in the right or left eye of each study participant using the Dynamic Vessel Analyzer (DVA, IMEDOS Systems, Jena, Germany). Units of measure mm, reported as a %change from baseline, before and after treatment.
Change in neuronal activity | 1 week
  EEG signal will be collected to generate spectral data. These data will be used for comparison of EEG activity between before and after treatment. Units of measure - power spectral density. Reported as a %change from baseline, before and after treatment.

SECONDARY OUTCOMES:
Change in microvascular endothelial function | 1 week
  Changes in microvascular endothelial function will be assessed using laser speckle contrast imaging (LSCI) in the hand using the flow mediated dilation approach. The change in skin perfusion is calculated and reported as a %change from baseline, between before and after treatment. Units of measure - perfusion index (arbitrary units). Reported as a %change from baseline, before and after treatment.
Change in macrovascular endothelial function | 1 week
  Changes in macrovascular endothelial function will be assessed using sonography during flow mediated dilation approach. The change in brachial artery diameter (mm) is calculated and reported as a %change from baseline, between before and after treatment.
Change in Glycocalyx - perfused boundary region | 1 week
  Video recordings of the sublingual vasculature will be performed using the high definition video camera GlycoCheck (Microvascular health solutions). Data collected will include perfused boundary region (um), and will be used for comparison before and after treatment.
Change in capillary density | 1 week
  Video recordings of the sublingual vasculature will be performed using the high definition video camera GlycoCheck (Microvascular health solutions). Data collected will include capillary density (mm/mm^2), and will be used for comparison before and after treatment.
Change in red blood cell velocity | 1 week
  Video recordings of the sublingual vasculature will be performed using the high definition video camera GlycoCheck (Microvascular health solutions). Data collected will include red blood cell velocity (um/sec), and will be used for comparison before and after treatment.
Change in grip strength | 1 week
  The change in hand grip strength will be measured before and after intervention. Data collected will include measurements of power in kg for left and right hand respectively
Change in Attention | 1 week
  CANTAB research attention test.Reported as a %change from baseline, before and after treatment.
Change in Working Memory | 1 week
  CANTAB research working memory test.Reported as a %change from baseline, before and after treatment.
Change in Executive Function | 1 week
  CANTAB research executive function test.Reported as a %change from baseline, before and after treatment.
Change in Processing Speed | 1 week
  CANTAB research processing speed test.Reported as a %change from baseline, before and after treatment.
Blood collection | 1 week
  Blood samples will be collected to measure L-Citrullin related metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Andriy Yabluchanskiy, MD, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Andriy Yabluchanskiy, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
PhysioNet